CLINICAL TRIAL: NCT06309992
Title: Multicentre, Randomised, Double-blind, Placebo-controlled, 48-week, Phase III Trial to Evaluate the Efficacy and Safety of Survodutide Administered Subcutaneously in Participants With Overweight or Obesity and Presumed or Confirmed Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study to Test Whether Survodutide Helps People Living With Obesity or Overweight and With a Confirmed or Presumed Liver Disease Called Non-alcoholic Steatohepatitis (NASH) to Reduce Liver Fat and to Lose Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0056; 2023-505303-23-00 (Registry Identifier: CTIS); U1111-1299-9925 (Registry Identifier: WHO registry)
Record Dates: First submitted 2024-03-08; First posted 2024-03-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Non-Alcoholic SteatoHepatitis (NASH)
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental)
  Interventions: Drug: Survodutide
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Survodutide — Survodutide
  Arms: Treatment arm
Drug: Placebo — Placebo matching survodutide
  Arms: Placebo arm

SUMMARY:
This study is open to adults who are at least 18 years old and have

* presumed or confirmed NASH together with overweight or obesity and
* a body mass index (BMI) of 30 kg/m² or more, or
* a BMI of 27 kg/m² and at least one weight-related health problem.

People with a history of other chronic liver diseases cannot take part in this study.

The purpose of this study is to find out whether a medicine called survodutide helps people living with obesity or overweight and a confirmed or presumed liver disease called nonalcoholic steatohepatitis (NASH) to have less liver fat and to lose weight. Participants are put into 2 groups randomly, which means by chance. 1 group gets different doses of survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Every participant has a 2 in 3 chance of getting survodutide. Participants and doctors do not know who is in which group. Participants inject survodutide or placebo under their skin once a week for about 1 year. In addition to the study medicine, all participants receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for about 1 year and 3 months. During this time, it is planned that participants visit the study site up to 14 times and receive 3 phone calls by the site staff. The doctors check participants' health and take note of any unwanted effects. The participants' body weight is regularly measured. At 3 of the visits, the participants' liver is measured using different imaging methods. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Key inclusion criteria:

* Age ≥18 years at the time of signing informed consent, and at least the legal age of consent in countries where it is >18 years
* BMI ≥30 kg/m², OR BMI ≥27 kg/m² and at least one of the following weight-related comorbidities at screening:

  * Hypertension (defined as repeated, i.e. at least 3 measurements in resting condition, Systolic Blood Pressure (SBP) values of ≥140 mmHg and/or Diastolic Blood Pressure (DBP) values of ≥90 mmHg in the absence of anti-hypertensive treatment, or intake of at least 1 antihypertensive drug to maintain a normotensive blood pressure)
  * Dyslipidaemia (defined as at least 1 lipid-lowering treatment required to maintain normal blood lipid levels, or lowdensity lipoprotein (LDL) cholesterol ≥160 mg/dL (≥4.1 mmol/L) or triglycerides ≥150 mg/dL (≥1.7 mmol/L), or high-density lipoprotein (HDL) cholesterol <40 mg/dL (<1.0 mmol/L) for men or HDL cholesterol <50 mg/dL (<1.3 mmol/L) for women
  * Obstructive sleep apnoea
  * Cardiovascular disease (e.g. heart failure with New York Heart Association (NYHA) functional class II-III, history of ischaemic or haemorrhagic stroke or cerebrovascular revascularisation procedure [e.g. carotid endarterectomy and/or stent], MI, coronary artery disease, or peripheral vascular disease)
  * Type 2 diabetes mellitus (T2DM) (diagnosed at least 180 days prior to screening, with glycated haemoglobin [HbA1c] ≥6.5% (48 mmol/mol) and <10% (86 mmol/mol) as measured by the central laboratory at screening)
* History of at least one self-reported unsuccessful dietary effort to lose body weight Further inclusion criteria apply.

Key exclusion criteria:

* Current or history of significant alcohol consumption (defined as intake of >210 g/week in men and >140 g/week in women on average over a consecutive period of more than 3 months) or inability to reliably quantify alcohol consumption based on the investigator's judgement within the last 5 years.
* Intake of medications associated with liver injury, hepatic steatosis or steatohepatitis.
* History of other chronic liver diseases (e.g. viral hepatitis, autoimmune liver disease, primary biliary cholangitis , primary sclerosing cholangitis, Wilson's disease, hemochromatosis, Alpha-1 Antitrypsin (A1At) deficiency, history of liver transplantation). Hepatitis B and C testing will be done at Visit 1. Participants with positive hepatitis B surface antigen (HBsAg) should be excluded. Participants treated for hepatitis C must have a negative ribonucleic acid (RNA) test at screening and also be Hepatitis C virus (HCV) RNA negative for at least 3 years prior to screening in order to be eligible for the trial. Trial participants with positive HCV antibody and no history of HCV treatment require a negative HCV RNA test at screening to be eligible for the trial.
* Cirrhosis based on clinical assessment, abdominal imaging, liver histology or non-invasive tests assessed at screening (enhanced liver fibrosis (ELF) ≥11.3 or Fibrosis (FIB)-4 ≥3.48 or FibroScan® VCTE™ ≥20 kPa or MRE ≥4.68 kPa) or a history of cirrhosis.
* Current decompensated liver disease or previous hepatic decompensation (ascites, spontaneous bacterial peritonitis, portal hypertension bleeding, hepatic encephalopathy, hepatorenal syndrome).
* Evidence of portal hypertension (e.g. splenomegaly, oesophageal varices, or other portosystemic collateral pathways).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Relative reduction in liver fat content of at least 30% from baseline to Week 48 (yes/no) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) [%] | at baseline, at week 48
Relative change (%) in body weight [kg] from baseline to Week 48 | at baseline, at week 48

SECONDARY OUTCOMES:
Absolute change from baseline to Week 48 in liver fat content assessed by MRI-PDFF [%] | at baseline, at week 48
Relative change (%) from baseline to Week 48 in liver fat content assessed by MRI-PDFF [%] | at baseline, at week 48
Reduction from baseline to Week 48 in Iron corrected T1 (cT1) [ms] levels of ≥80 ms (yes/no) | at baseline, at week 48
Absolute change from baseline to Week 48 in alanine amino transferase (ALT) [U/L] levels | at baseline, at week 48
Relative change from baseline to Week 48 in alanine amino transferase (ALT) [U/L] levels | at baseline, at week 48
Absolute change from baseline to Week 48 in waist circumference [cm] | at baseline, at week 48
Relative change from baseline to Week 48 in waist circumference [cm] | at baseline, at week 48
Absolute change from baseline to Week 48 in Homeostasis Model Assessment -Insulin Resistance (HOMA-IR) (Fasting Plasma Insulin (FPI) [mlU/L] · Fasting Plasma Glucose (FPG) [mmol/L]/22.5) | at baseline, at week 48
Relative change from baseline to Week 48 in HOMA-IR (FPI [mlU/L] · FPG [mmol/L]/22.5) | at baseline, at week 48
Absolute change from baseline to Week 48 in liver stiffness [kPa] assessed by magnetic resonance elastography (MRE) | at baseline, at week 48
Relative change from baseline to Week 48 in liver stiffness [kPa] assessed by magnetic resonance elastography (MRE) | at baseline, at week 48
Absolute change in liver volume [mL] from baseline to Week 48 measured using MRI | at baseline, at week 48
Relative change in liver volume [mL] from baseline to Week 48 measured using MRI | at baseline, at week 48

CONTACTS AND LOCATIONS:
Locations (37):
- United States (33):
  - ARK Clinical Research, Fountain Valley, California
  - Velocity Clinical Research-Gardena-69773, Gardena, California
  - ARK Clinical Research, Long Beach, California
  - Catalina Research Institute, LLC - Montclair, Montclair, California
  - Velocity Clinical Research-North Hollywood-69852, North Hollywood, California
  - Velocity Clinical Research-Panorama City-68861, Panorama City, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Segal Drug Trials, Delray Beach, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Covenant Metabolic Specialists, LLC - Fort Myers, Fort Myers, Florida
  - Velocity Clinical Research-Hallandale Beach-67888, Hallandale, Florida
  - Nature Coast Clinical Research-Inverness-48221, Inverness, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Verus Clinical Research Corporation, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Covenant Research and Clinics, LLC, Sarasota, Florida
  - Springfield Clinic, LLP, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas Medical Clinic PA, Topeka, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - DSI Research Northridge LLC, Dayton, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Velocity Clinical Research, Austin, Austin, Texas
  - Amel Med LLC, Georgetown, Texas
  - Gastroenterology and Liver Research LLC, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Accurate Clinical Research, Inc., Humble, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Velocity Clinical Research, Waco, Waco, Texas
  - GI Select Health Research LLC, Richmond, Virginia
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Younossi ZM, Razavi H, Sherman M, Allen AM, Anstee QM, Cusi K, Friedman SL, Lawitz E, Lazarus JV, Schuppan D, Romero-Gomez M, Schattenberg JM, Vos MB, Wong VW, Ratziu V, Hompesch M, Sanyal AJ, Loomba R. Addressing the High and Rising Global Burden of Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) and Metabolic Dysfunction-Associated Steatohepatitis (MASH): From the Growing Prevalence to Payors' Perspective. Aliment Pharmacol Ther. 2025 May;61(9):1467-1478. doi: 10.1111/apt.70020. Epub 2025 Feb 18. PMID 39967239
- See also: Related Info — https://www.mystudywindow.com